CLINICAL TRIAL: NCT02149459
Title: Improving the Response of Recurrent Glioma to Radiation Therapy Through Metabolic Intervention
Brief Title: Treatment of Recurrent Brain Tumors: Metabolic Manipulation Combined With Radiotherapy
Acronym: SMC 0712-13
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0712-YL-CTIL
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Brain Neoplasms
Keywords: Radiotherapy; Ketosis; Metformin; Magnetic Resonance Imaging; Metabolome; Insulin; recurrent brain tumors; gliomas; glioblastomas; astrocytomas
MeSH Terms: conditions — Brain Neoplasms; Ketosis; Insulin Resistance; Glioma; Glioblastoma; Astrocytoma | interventions — Radiotherapy; Metformin; Hypoglycemic Agents; Biguanides; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment arm (Experimental): Partial brain re-irradiation combined with metabolic intervention (low carbohydrate diet and/or metformin treatment)
  Interventions: Radiation: Partial brain re-irradiation.; Drug: Metformin; Behavioral: low carbohydrate diet

INTERVENTIONS:
Radiation: Partial brain re-irradiation. — Partial brain re-irradiation to a dose of 30-35Gy delivered over 2 weeks (10 fractions).
  Other Names: radiotherapy; radiation therapy (RT); fractionated stereotactic radiation (FSR); hypo-fractionated radiation therapy
Drug: Metformin — Different cohorts will receive no, low dose or higher dose metformin.
  Other Names: glucophage; antidiabetic drug; biguanide
Behavioral: low carbohydrate diet — Under close supervision of a dietician, patients will receive a low carbohydrate diet, enriched as necessary with medium chain triglyceride (MCT) supplements.

SUMMARY:
Recurrent brain tumours are extremely aggressive and despite optimal treatment, median survival is less than two years. One of the standard treatment options in this situation is radiation therapy. Currently there is intense scientific interest concerning the abnormal energy metabolism in cancer cells. All cells require energy in order to function, obtaining 'fuel' molecules such as glucose and fatty acids from the blood stream. Brain tumours exhibit "metabolic reprogramming", meaning that their energy requirements and utilization of fuel molecules are quite different from normal cells. Brain tumour cells are exquisitely dependant on glucose as a source of energy. Animal studies have shown that when these tumours are deprived of glucose they are very sensitive to radiation therapy.

In this clinical trial the investigators combine radiation therapy with a low-carbohydrate diet, in patients with recurrent brain tumours. In addition, subjects will receive medication with metformin, a drug usually used to treat diabetes. Metformin inhibits glucose metabolism within cancer cells, and additionally has reported intrinsic anti-cancer activity. Subjects will undergo advanced imaging and hormonal studies before, during and after the trial in order to obtain maximal translational-scientific impact.

The hypothesis:

The metabolic changes induced by the combination of a moderately-low carbohydrate diet combined with supplementary MCT and metformin therapy will selectively starve tumor cells. While normal brain cells are capable of deriving energy from ketone bodies during glucose restriction, tumor cells remain largely glucose-dependent for energy due to oncogene induced down-regulation of oxidative phosphorylation. While the tumor cells are in this 'vulnerable' state they will be less able to repair the damage induced by ionizing radiation.

Short-term implementation of the metabolic intervention (i.e. combined diet and metformin therapy) prior to, during, and after hypofractionated (2 week) radiation therapy is expected to increase tolerability, increase compliance and avoid the chronic metabolic complications associated with extreme carbohydrate restriction diets.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to participate in diet/metformin intervention for the 8 week period.
* Patients must have a previously histologically or cytologically confirmed glioma (astrocytic or oligodendroglial supratentorial tumors grades 2, 3 or 4 according to the WHO 2007 classification 82) that has been previously treated with fractionated radiation therapy and now shows evidence of recurrence. There is no limit regarding the number / type of previous therapies that the patient has received for glioma, aside from exceptions mentioned below. If the brain tumor is in an eloquent location (e.g. brain stem) a clinical diagnosis is sufficient.
* Patients must have recovered from the toxic effects of prior therapy.
* Patients must have recovered from the effects of any prior surgery to any part of the body. There must be a minimum of 10 days from the day of surgery to the day of registration. For core or needle biopsy, a minimum of 7 days must have elapsed prior to registration.
* Patients may have previously undergone more than one craniotomy.
* Prior treatment with cytotoxic and biological agents is permissible. There should be at least a 2 week break between prior treatment and enrollment.
* Prior treatment with fractionated radiation therapy (up to 66Gy) is an eligibility criterion, however this should have been completed ≥ 4 weeks prior to enrollment.
* One prior single fraction radio-surgical procedure within the treatment field is acceptable if V12<5cc (V12 is the volume of brain receiving 12 or more Gy). Additional radio-surgical procedures outside of the treatment area are acceptable.
* Age >=18 years.
* ECOG performance status <2 (Karnofsky>60%).
* Life expectancy of greater than 2 months.
* Patients must have normal organ and marrow function as defined below:

  * -leukocytes >2,000/mcL
  * -absolute neutrophil count >1,200/mcL
  * -platelets >80,000/mcL
  * -AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
* No contra-indications of metformin use:

  * Metformin allergy
  * Renal failure, creatinine levels over 150 μmol/l (1.7 mg/dL)
  * Liver disease
  * Current alcohol abuse
* Women of childbearing potential must have a negative β-HCG pregnancy test documented within 14 days of registration.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known to suffer from one of the following metabolic disorders (all rare):

  * Carnitine deficiency (primary)
  * Carnitine palmitoyltransferase (CPT) I or II deficiency
  * Carnitine translocase deficiency
  * β-oxidation defects
  * Medium-chain acyldehydrogenase deficiency (MCAD)
  * Long-chain acyl dehydrogenase deficiency (LCAD)
  * Short-chain acyl dehydrogenase deficiency (SCAD)
  * Long-chain 3-hydroxyacyl-CoA deficiency
  * Medium-chain 3-hydroxyacyl-CoA deficiency.
  * Pyruvate carboxylase deficiency
  * Porphyria
* Patients receiving insulin or oral medication on a daily basis for diabetes mellitus
* Known severe dyslipidemia: total cholesterol >400 mg/dl, LDL cholesterol > 300 mg/dl, triglycerides > 500 mg/dl
* Contraindications to metformin use:

  * Metformin allergy
  * Renal failure: creatinine levels over 150 μmol/l (1.7 mg/dL)
  * Liver disease
  * Current alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 8 weeks
  The investigators will track adverse events in order to determine the safety of the intervention.
Number of patients completing the trial. | 8 weeks
  We will track patient compliance in order to determine the tolerability of the intervention.

SECONDARY OUTCOMES:
Number of patients whose brain tumors respond on imaging. | 8 weeks
Number of patients who demonstrate changes in systemic energy metabolism. | 8 weeks
  We will assess plasma levels of glucose, insulin and other relevant hormones before, during and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yaacov R Lawrence, MA MBBS MRCP, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel